CLINICAL TRIAL: NCT03045393
Title: Pilot Study of Mirvetuximab Soravtansine (IMGN853) in Folate Receptor Alpha (FRα)-Expressing, Triple Negative Breast Cancer (TNBC) With Residual Disease Post Standard Neoadjuvant Chemotherapy
Brief Title: Mirvetuximab Soravtansine (IMG853) in Folate Receptor Alpha-expressing TNBC
Acronym: IMGN853
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Inadequate enrollment
Sponsor: Duke University (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00074621
Record Dates: First submitted 2017-02-03; First posted 2017-02-07 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer Triple Negative
Keywords: Neoadjuvant; Breast Cancer; Folate Receptor Alpha; FRa; TNBC; Triple Negative Breast Cancer; Preoperative; Presurgery; Mirvetuximab Soravtansine; IMGN853
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — mirvetuximab soravtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mirvetuximab Soravtansine (Experimental): Participants will receive 2 doses of Mirvetuximab Soravtansine after neoadjuvant chemotherapy and before surgical resection of tumor.
  Interventions: Drug: Mirvetuximab Soravtansine (IMGN853)

INTERVENTIONS:
Drug: Mirvetuximab Soravtansine (IMGN853) — Mirvetuximab Soravtansine is a targeted drug for tumors that express high levels of folate receptor alpha.

SUMMARY:
The main purpose of this study is to determine how 2 doses mirvetuximab soravtansine affects the amount and activity of folate receptor alpha proteins in tumor cells of patients who have completed standard neoadjuvant treatment and are scheduled to have their tumors surgically removed.

DETAILED DESCRIPTION:
The folate receptor alpha protein is important in tumor growth and can be over-expressed in some tumor cells. The word "over-expressed" in this situation means that there are too many copies of the protein on the surface of the cell when compared to a healthy, normal cell, and this helps the tumor continue to grow in size. Mirvetuximab soravtansine acts by targeting the folate receptor in tumor cells. In animal models, mirvetuximab soravtansine is highly effective in decreasing tumor size. This suggests that mirvetuximab soravtansine may help shrink or stop growth of folate receptor alpha positive breast cancer in this study.

In this study the investigator will be looking at how folate receptor alpha expression changes following 2 doses of neoadjuvant mirvetuximab soravtansine. The investigator will also look to evaluate the safety of this regimen, measure any change in tumor size, associate folate receptor alpha expression with a change in tumor size, and describe any changes in Ki-67 and percent of apoptotic cells in this population.

ELIGIBILITY:
Screening Inclusion Criteria:

* Signed informed screening consent form with HIPAA authorization for release of personal health information.
* Research personnel will review medical records of subjects consenting to screening to ensure no obvious factors would exclude them from the treatment portion of the study (e.g., history of cirrhosis of the liver) and to confirm diagnosis and staging
* Histological confirmation of triple negative breast cancer (TNBC) biopsy report
* Stage 1-3 tumors > 1cm in maximal diameter.
* Standard neoadjuvant chemotherapy NAC and definitive surgery planned (NOTE: NAC chemotherapy will be per standard of care, and not dictated by this clinical trial)
* Must be able to supple sufficient tissue (block or slides) from diagnostic biopsy to undergo testing.

Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information.
* Must have operable tumor ≥ 1cm determined by and obtained less than 9 weeks after completion of standard NAC
* Must be able to meet study schedule: 2 doses of mirvetuximab soravtansine administered 3 weeks apart and surgery within 9 weeks of last dose of NAC.
* Willing to undergo biopsy for research purposes only (before and after), and to allow surgical tissue sample from surgery to be used for research purposes
* May have symptoms however must be ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work)
* Demonstrate adequate organ function through labs
* Females of childbearing years must have a negative serum pregnancy test within 48 hours prior to dose 1 mirvetuximab soravtansine. NOTE: Sexually mature females are considered of child bearing potential unless they are surgically sterile (have undergone a hysterectomy, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months
* Females of childbearing potential must be willing to abstain from heterosexual activity or to use two effective methods of contraception from the time of informed consent until 4 months after the last dose of mirvetuximab soravtansine

Exclusion Criteria:

* Pregnant or breastfeeding, or plan to be pregnant within projected duration of the trial. (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
* Has a known additional malignancy that is active and/or progressive requiring treatment within 3 years of first dose.
* Prior treatment with mirvetuximab soravtansine
* Treatment with any investigational drug within 6 weeks of first clinical dose
* Subjects with > Grade 1 peripheral neuropathy
* Active or chronic corneal disorder, including but not limited to the following:

  * Sjogren's syndrome
  * Fuchs corneal dystrophy (requiring treatment)
  * History of corneal transplantation
  * Active herpetic keratitis
  * Active ocular conditions requiring on-going treatment/monitoring such as wet age-related macular degeneration requiring intravitreal injections, active diabetic retinopathy with macular edema, presence of papilledema, and acquired monocular vision.
* Serious concurrent illness or clinically-relevant active infection
* Cytomegalovirus infection
* Any concurrent infectious disease, requiring IV antibiotics within 2 weeks of first dose of mirvetuximab soravtansine
* Significant cardiac disease including
* History of neurological conditions that would confound assessment of treatment-emergent neuropathy other than ≤ Grade 1 peripheral neuropathy including multiple sclerosis or other demyelinating disease and/or eaton-lambert syndrome (para-neoplastic syndrome)" Diabetes is allowed.
* History of hemorrhagic or ischemic stroke within 6 months prior to first dose of mirvetuximab soravtansine
* History of cirrhotic liver disease
* Previous clinical diagnosis of non-infectious pneumonitis or non-infectious interstitial lung disease
* Prior hypersensitivity to monoclonal antibodies
* History or evidence of thrombotic or hemorrhagic disorders within 6 months prior to first dose of mirvetuximab soravtansine
* Required used of folate-containing supplements (e.g. for folate deficiency)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Change in breast tumor FRα expression before and after treatment with mirvetuximab soravtansine | Baseline up to 9 weeks
  Assessed by immunohistochemistry (IHC) (1) after completion of neoadjuvant chemotherapy, prior to treatment with mirvetuximab soravtansine; (2) at definitive surgery, after treatment with mirvetuximab soravtansine and scored (0 = no receptors, 1 = small number of receptors, 2 = medium number of receptors, 3 = large number of receptors).

SECONDARY OUTCOMES:
Change in breast tumor FRα expression before and after neoadjuvant chemotherapy | Baseline up to 9 weeks
  Assessed by immunohistochemistry (IHC) (1) at initial cancer diagnosis, prior to initiation of neoadjuvant chemotherapy; (2) after completion of neoadjuvant chemotherapy and scored (0 = no receptors, 1 = small number of receptors, 2 = medium number of receptors, 3 = large number of receptors).
Total number of grade 3 and 4 toxicities | Baseline up to 9 weeks
  Graded via NCI CTCAE v4.03
Number of treatment-emergent adverse events (TEAEs) precluding second dose | Baseline up to 9 weeks
  Assessed by the number of subjects that cannot receive the second dose of mirvetuximab soravtansine
Number of treatment-emergent adverse events (TEAEs) delaying surgery | Baseline up to 9 weeks
  Assessed by the number of subjects that have surgery delayed past 9 weeks due to TEAE
Total number of partial or complete responses | Baseline up to 9 weeks
  Evaluated by the number of subjects that have either a partial or complete radiologic response by 2D ultrasound. (Partial response = reduction of the largest unidimensional tumor measurement of >30%; Complete response = no evidence of tumor remaining)
Change in tumor cell proliferation, as measured by Ki67 expression | Baseline up to 9 weeks
  Changes in Ki67 expression will be measured before and after 2 doses of mirvetuximab soravtansine.
Change in tumor cell death markers | Baseline up to 9 weeks
  Changes in apoptotic markers will be measured before and after 2 doses of mirvetuximab soravtansine.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Blackwell, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States